CLINICAL TRIAL: NCT00917488
Title: Glycyphagus Domesticus Allergen Extract. Determination of the in Vivo Biological Activity in Histamine Equivalent Units (HEP).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: María José Gómez / Clinical Development Manager, Laboratorios LETI S.L.Unipersonal
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 108-PR-PRI-147; 2007-000904-33 (EudraCT Number)
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic
Keywords: Allergen extract Standardization
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Four concentrations of Glycyphagus domesticus allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, was tested in every patient in duplicate on the volar surface of the forearm.
  Interventions: Other: Standardization of allergenic extract (Gly. domesticus)

INTERVENTIONS:
Other: Standardization of allergenic extract (Gly. domesticus) — Allergenic extract for cutaneous prick-test

SUMMARY:
The main purpose of the trial is to prove the therapeutic value of the product and enable an effective and safe dosage schedule to be recommended

DETAILED DESCRIPTION:
The objective of this study is to determine the biologic activity of a Glycyphagus domesticus allergen extract in histamine equivalent prick (HEP) units, in order to be used as in-house reference preparation (IHRP).

The skin testing procedure, based on the Nordic Guidelines is the reference method for the biological calibration of in-House Reference Preparations (IHRP). The method is not intended for routine testing of allergen extracts. The use of this procedure is the basis for the definition of biological activity units: "the activity of an allergen extract is 10,000 Biological Units (BU) per ml (10 HEP per ml), when the extract provokes an specific skin reaction in the median sensitive patient with a wheal of the same size as a wheal provoked by a positive reference solution consisting of histamine 54.3 mmol/l (for example histamine dihydrochloride 10 mg/ml), when both solutions are administrated using the same technique (prick testing) on at least 20 individuals who are clinically allergic and cutaneously reactive to the allergen concerned".

ELIGIBILITY:
Subject inclusion criteria:

1. A documented positive case history with inhalation allergy (rhinitis and/or rhinoconjunctivitis and/or asthma) related to Glycyphagus domesticus.
2. Positive skin prick test with an available preparation of the same allergen extract (a wheal major diameter of at least 3 mm) and/or a positive test for specific IgE.
3. Mean of the areas of the wheals provoked by histamine dihydrochloride (10 mg/ml) ≥ 7 mm2.
4. Age ≥ 18 years and ≤ 50 years
5. Subject can be male or female
6. Subject must be capable of providing written informed consent

Subject exclusion criteria:

1. Subjects should not be excluded due to low or high sensitivity to Glycyphagus domesticus.
2. Immunotherapy in the past 2 years with an allergen preparation known to interfere with the allergens to be tested.
3. Use of drugs that may interfere with the skin reactions.
4. Pregnancy, dermographism, atopic dermatitis (locally at the test site), urticaria.
5. Any disease which prohibits the use of adrenaline (hyperthyroidism, arterial hypertension, cardiopathy, etc.)
6. Lack of cooperation which may interfere with the study, or subjects with severe psychiatric, psychological or neurological disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Wheal size area (mm2) on the skin at the site of the puncture during the immediate phase. | 45 minutes per subject

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Moreno, MD, PhD, Principal Investigator
Locations (1):
- Clinica Dr. Lobatón, Cadiz, Cadiz, Spain